CLINICAL TRIAL: NCT00634270
Title: A Phase II Study of the mTOR Inhibitor Sirolimus in Neurofibromatosis Type 1 Related Plexiform Neurofibromas
Acronym: Protocol 102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's National Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); National Cancer Institute (NCI) (NIH); University of Chicago (Other); University of Utah (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F071019012; DOD: W81XWH-05-615. (Other: Department of Defense); UAB: 251558. (Other: UAB Link Number)
Record Dates: First submitted 2008-02-20; First posted 2008-03-13 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Neurofibromatosis Type 1
Keywords: Plexiform, Neurofibromatosis Type 1, Sirolimus, Phase II
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Design
  * Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing.
  * Disease status will be evaluated using volumetric MRI analysis at regular intervals.
  * The plasma pharmacokinetics and pharmacodynamics of sirolimus will be evaluated, as will pharmacogenetic polymorphisms and their influence on the metabolism of sirolimus in this patient population.
  * Pain reduction and quality of life outcomes will also be assessed.
  * Toxicity of chronic sirolimus administered will be evaluated using physical and laboratory evaluations.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — This phase II study will evaluate children and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with sirolimus. It is divided in two strata. The first stratum will evaluate time to progression (TTP) in children and adults with NF1 and progressive plexiform neurofibromas with the potential to cause significant morbidity treated with sirolimus. The second stratum will evaluate objective radiographic response to sirolimus in children and adults with NF1 and inoperable plexiform neurofibromas with the potential to cause significant morbidity that do not have documented progression of the PN at time of trial entry.
  Other Names: Rapamune; Rapamycin

SUMMARY:
Treatment Overview

This phase II study will evaluate the activity of sirolimus in children and adults with NF1 and inoperable plexiform neurofibromas that have the potential to cause significant morbidity. The following disease strata will be studied:

Stratum 1: Progressive plexiform neurofibroma(s) that have the potential to cause significant morbidity. The endpoint will be time to tumor progression based on volumetric tumor measurements.

Stratum 2: Plexiform neurofibromas without documented radiographic progression at trial entry. The endpoint will be radiographic response. As of May 2009, Stratum 2 was closed to enrollment. Stratum 1 is active.

DETAILED DESCRIPTION:
ABSTRACT/SCHEMA

Sirolimus will be provided as oral solution 1 mg/ml to allow for precise dose adjustments. The tablet and oral solution forms are clinically equivalent (2003). Sirolimus will be administered orally twice daily (approximately every 12 hours) for a 28 day course with no rest period between courses. Sirolimus should be taken by the patient consistently either with or without food. Sirolimus should NOT be taken with grapefruit juice or with other effectors of CYP3A4 (see section 4.1.7). Dietary habits around the time of sirolimus intake should be as consistent as possible throughout the study, and in particular, during those periods when samples are being taken for pharmacokinetic analyses (if applicable). Limited exposure to sunlight and wearing sunscreen is recommended while taking this drug. If you miss a dose, treatment should continue without making up the missed dose.

The starting dose will be 0.8 mg/m2 BSA per dose. Each patient's dose will be rounded to the nearest 0.1 mg (adult average 1.6 mg per dose). The BSA should be calculated based on an accurate height and weight measurement performed according to institutional guidelines, or using the following formula:

Square root of: (Height[cm] X Weight[kg]/3,600)

Dosing will be pharmacokinetically adjusted to maintain trough sirolimus levels within the target range of 10-15 ng/ml. (Appendix IV-A). The first sirolimus level will not be measured until week 2 to allow for loading to occur and to approach steady state concentrations. If patients are unable to achieve target trough sirolimus levels within 4 weeks, patients may be asked to have mini-pharmacokinetics of 3 blood draws, in addition to a trough level, in order to better estimate patient's dose. The extra trough sirolimus levels will be at: 1 hour, 3 hours, and 4-6 hours after a sirolimus dose.

Sirolimus doses will be adjusted pharmacokinetically and will account for changes in body surface area.

Dose modifications for patients who experience toxicities are outlined in Section 8.0.

Sirolimus should be re-taken if vomiting occurs within 15 minutes of taking the dose, but not if vomiting occurs more than 15 minutes after taking sirolimus. Patients or their parents/guardians will keep a diary to document the intake of each dose of sirolimus and potential side effects. The patient diary should be reviewed with the patient's family at each required clinical study evaluation. In addition, leftover study medication should be collected at each on study evaluation, and drug should be accounted for at this time (Appendix V).

A treatment course will consist of 4 weeks of therapy. For stratum 1 treatment may continue until disease progression or unacceptable toxicity occurs. Patients entered on stratum 2 may receive up to a maximum of 6 courses (i.e. 24 weeks) of therapy unless there is evidence of objective radiographic response, as defined in Section 13.0 (> to 20% decrease in PN volume), tumor progression, or unacceptable toxicity. Patients who experience unacceptable toxicity or disease progression will be removed from treatment with sirolimus. Patients with documented radiographic response may continue treatment with sirolimus for up to 6 treatment courses after the maximum response.

Background

* Patients with Neurofibromatosis 1 (NF1) have an increased risk of developing tumors of the central and peripheral nervous system, including plexiform neurofibromas (PN), which are benign nerve sheath tumors that are among the most debilitating complications of NF1. Plexiform neurofibromas appear to have the fastest growth rate in young children. There are no standard treatment options for PN other than surgery, which is often difficult due to the extensive growth and invasion of surrounding tissues.
* Mammalian Target of rapamycin (mTOR), a serine/threonine kinase regulated by the phosphoinositol 3 kinase (PI3K), acts as a master switch of cellular catabolism and anabolism and controls protein translation, angiogenesis, cell motility, and proliferation.
* The NF1 tumor suppressor, neurofibromin, regulates the mTOR pathway activity, with increased mTOR activation observed in NF1-deficient cells and tumors from NF1 patients.
* Sirolimus is a macrolide antibiotic that inhibits mTOR activity, preventing phosphorylation (and activation) of p70S6K, 4E-BP1, and other proteins involved in cell motility, angiogenesis, and cell growth control.

Primary Objectives

• To determine whether the mTOR inhibitor sirolimus, administered using pharmacokinetically-guided dosing: Increases time to disease progression based on volumetric MRI measurements in children and adults with neurofibromatosis type 1 (NF1) and progressive plexiform neurofibromas (PN).

Results in objective radiographic responses based on volumetric MRI measurements in children and adults with NF1 and inoperable PN in the absence of documented radiographic progression at trial entry.

* To evaluate the feasibility and toxicity of chronic sirolimus administration in this patient population.
* To characterize the pharmacokinetic profile (profile includes pharmacodynamics and pharmacogenetics) of sirolimus when administered to this patient population.

Eligibility

* Patients ≥ 3 years old with NF1 AND
* Inoperable, measurable, radiographically PROGRESSIVE PN that have the potential to cause significant morbidity.

OR

• Inoperable, measurable PN WITHOUT documented progression that have the potential to cause significant morbidity.

Design

* Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing.
* Disease status will be evaluated using volumetric MRI analysis at regular intervals.
* The plasma pharmacokinetics and pharmacodynamics of sirolimus will be evaluated, as will pharmacogenetic polymorphisms and their influence on the metabolism of sirolimus in this patient population.
* Pain reduction and quality of life outcomes will also be assessed.
* Toxicity of chronic sirolimus administered will be evaluated using physical and laboratory evaluations.

EXPERIMENTAL DESIGN SCHEMA

GOALS AND OBJECTIVES (SCIENTIFIC AIMS)

Primary Aims

To determine whether the mTOR inhibitor sirolimus, administered orally twice daily on a continuous dosing schedule (1 course = 28 days) using pharmacokinetically-guided dosing:

Increases time to disease progression based on volumetric MRI measurements in children and young adults with neurofibromatosis type 1 (NF1) and inoperable progressive plexiform neurofibromas (PN),

To evaluate the feasibility and toxicity of chronic sirolimus administration in this patient population.

To characterize the pharmacokinetic profile of sirolimus when administered to this patient population.

Secondary Aims

To evaluate quality of life during treatment with sirolimus and to assess preliminary correlations of response with quality-of-life outcomes.

To evaluate the effect of sirolimus on clinical response by reduction in pain, or improvement in function or performance scale.

ELIGIBILITY:
Inclusion Criteria: all patients (stratum 1 and 2):

* All patients must have the clinical diagnosis of NF1 using the NIH Consensus Conference criteria.
* Six or more café-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects).
* Freckling in the axilla or groin.
* Optic glioma.
* Two or more Lisch nodules.
* A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex).
* A first-degree relative with NF1.
* Patients must have plexiform neurofibroma(s) that have the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or significant cosmetic problems, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Patients with paraspinal plexiform neurofibromas will be eligible for this trial. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings, but should be considered if malignant degeneration of a plexiform neurofibroma is clinically suspected.
* Age: Patients must be greater than or equal to 3 years of age at the time of study entry.
* Durable Power of Attorney: Adults evaluated for this study will be offered a durable power of attorney. Adults who are unable to provide informed consent will have to have a durable power of attorney in order to participate in this trial.
* Disease status: Measurable disease: Patients must have measurable plexiform neurofibroma(s) amenable to volumetric MRI analysis. For the purpose of this study, a measurable lesion will be defined as a lesion of at least 3 cm measured in one dimension.
* Performance Level: Karnofsky greater than or equal to 50% for patients > 10 years of age and Lansky greater than or equal to 50 for patients less than or equal to 10 years of age (Appendix IV). Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy: Patients who underwent surgery for a progressive plexiform neurofibroma will be eligible to enter the study after the surgery, provided the plexiform neurofibroma was incompletely resected and is measurable. Patients are only eligible if complete resection of a plexiform neurofibroma with acceptable morbidity is not feasible, or if a patient with surgical option refuses surgery. Patients may have been previously treated for a plexiform neurofibroma but must have fully recovered from the acute toxic effects of all prior chemotherapy or radiotherapy prior to entering this study.
* a. Myelosuppressive chemotherapy: Must not have received within 4 weeks of entry onto this study.
* b. Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor that supports platelet, red or white cell number or function.
* c. Biologic (anti-neoplastic agent): At least 14 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur. These patients must be discussed with the Study Chair on a case-by-case basis.
* d. Investigational Drugs: Patients must not have received an investigational drug within 4 weeks.
* e. Steroids: Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* f. CYP3A4 inhibitors: Patients may not be currently receiving strong inhibitors of CYP3A4, and may not have received these medications within 1 week of entry. These include: Macrolide Antibiotics: clarithromycin, telithromycin, erythromycin, troleandomycin; Gastrointestinal prokinetic agents: cisapride, metoclopramide; Antifungals: itraconazole, ketoconazole, fluconazole, voriconazole, clotrimazole; Calcium channel blockers: verapamil, diltiazem, nicardipine; and, Other drugs: rifampin, bromocriptine, cimetidine, danazol, cyclosporine oral solution.
* Grapefruit juice.
* g. CYP3A4 inducers: Patients must also avoid strong inducers of CYP3A4 and may not have received these medications within 1 week of entry. These include: Anticonvulsants: carbamazepine, phenobarbital, phenytoin; Antibiotics: rifabutin, rifapentine; Herbal preparations: St. John's wort (Hypericum perforatum, hypericine).
* h. Enzyme inducing anticonvulsants : Patients may not be taking enzyme - inducing anticonvulsants, and may not have received these medications within 1 week of entry, as these patients may experience different drug disposition. These medications include: Carbamazepine (Tegretol), Felbamate (Felbtol), Phenobarbitol, Phenytoin (Dilantin), Primidone (Mysoline), Oxcarbazepine (Trileptal), and, Herbal preparations: St. John's wort (Hypericum perforatum, hypericine).
* i. XRT: Greater than or equal to 6 months from involved field radiation to index plexiform neurofibroma(s); greater than or equal to 6 weeks must have elapsed if patient has received radiation to areas outside index plexiform neurofibroma(s).
* j. Surgery: At least 2 weeks since undergoing any major surgery.
* Organ Function Requirements; Adequate Bone Marrow Function Defined as: Peripheral absolute neutrophil count (ANC)greater than or equal to 1500/μL; Platelet count greater than or equal to 100,000/μL (transfusion independent); and Hemoglobin greater than or equal to 10.0 gm/dL (may receive RBC transfusions).
* Adequate Renal Function Defined as: A serum creatinine based on age, OR a creatinine clearance or radioisotope GFR greater than or equal to 70ml/min/1.73 m2
* Adequate Liver Function Defined As: Bilirubin (sum of conjugated + unconjugated) < or equal to 1.5 x upper limit of normal (ULN) for age, and SGPT (ALT)< or equal to 5 x upper limit of normal (ULN) for age, and Serum albumin > or equal to 2 g/dL.
* Fasting LDL Cholesterol: Patients must have a fasting LDL cholesterol of < 160 mg/dL; Patients taking a cholesterol lowering agent must be on a single medication and on a stable dose for at least 4 weeks

Specific eligibility criteria stratum 1 Disease status:

- Patients must have a progressive plexiform neurofibroma(s). Progression at the time of study entry is defined as: Presence of new plexiform neurofibromas on MRI or CT, OR A measurable increase of the plexiform neurofibroma (> or equal to 20% increase in the volume, or a > or equal to 13% increase in the product of the two longest perpendicular diameters, or a > or equal to 6% increase in the longest diameter) over the last two consecutive scans (MRI or CT), or over the time period of approximately one year prior to evaluation for this study.

Specific eligibility criteria stratum 2 Disease status:

- Radiographic disease progression as defined in Section 4.2.1 is not required for trial entry.

Exclusion Criteria:(Both Strata):

* Chronic treatment with systemic steroids or another immunosuppressive agent.
* Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Evidence of an active optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy. Patients not requiring treatment are eligible for this protocol.
* Dental braces or prosthesis that interfere with volumetric analysis of the neurofibroma(s).
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* A known history of HIV seropositivity or known immunodeficiency. HIV testing will not be required as part of this trial, unless HIV is clinically suspected.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sirolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A nasogastric tube (NG tube) is allowed.
* Women who are pregnant or breast feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the period they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Women of childbearing potential will be given a pregnancy test within 7 days prior to administration of sirolimus and must have a negative urine or serum pregnancy test.
* Patients who have received prior treatment with an mTOR inhibitor.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Patients who have an uncontrolled infection.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-04; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Korf, MD, Principal Investigator — The University of Alabama at Birmingham; Brian Weiss, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Roger Packer, MD, Study Director — Children's National Medical Center - Chairman of the NF Consortium
Locations (9):
- United States (9):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Existing and NF1 new patients at Consortium sites and partnering with the Children's Tumor Foundation.
Pre-assignment Details: Eligibility for Stratum 1 if evidence of progression and Stratum 2 if not evidence of progression.
Groups:
- Stratum 1: Design
  * Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing.
  * Disease status will be evaluated using volumetric MRI analysis at regular intervals.
  Sirolimus, Rapamycin: This phase II study will evaluate children and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with sirolimus. It is divided in two strata. The first stratum will evaluate time to progression (TTP) in children and adults with NF1 and progressive plexiform neurofibromas with the potential to cause sign
- Stratum 2: Non-randomized, single arm interventional strata for inoperable Plexiform Neurofibromas with potential to cause significant morbidity WITHOUT evidence of progression
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 49 (February 12, 2008) | 13
Completed | 46 | 12
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Of the 49 patients enrolled in Stratum 1; 46 were evaluable. Of the 13 enrolled in Stratum 2; 12 were evaluable. This information is also listed in the Analysis Population Descriptions and Additional Description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 49 | 13 | 62
Age, Continuous [Mean (Full Range); unit: years] | 9 [3 to 45] | 16 [3 to 35] | 10.46 [3 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 32
  Male | 25 | 5 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 35 | 10 | 45
  Unknown or Not Reports | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 49 | 13 | 62

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression Based on Volumetric MRI
Description: Median time to progression in Stratum 1 as defined as an increase of at least 20% of the volume of the primary lesion. Note: Since Stratum 2 looked at response rate only, median time to progression was not reviewed for this outcome.
Time Frame: 24 Months Stratum 1
Population: All evaluable participants. Note: In Stratum 2 the value was not assessed as "time to progression" therefore the appropriate response would be N/A. Stratum 2 was reported as response rate only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 46 | 0
Months | 15.4 [14.3 to 23.7] |

2. Primary Outcome: Results in Objective Radiographic Responses Based on Volumetric MRI Measurements in Children and Adults With NF1 and Inoperable PN in the Absence of Documented Radiographic Progression at Trial Entry
Description: Stratum 2 outcome - Response
Time Frame: 48 weeks Stratum 2
Population: Identify the index plexiform neurofibroma(s) for 3-D MRI evaluation based on prior imaging studies. The criteria for response was <20% increase in volume using RECIST v1.0. Response for 48 weeks was only assessed for Stratum 2.
Measure: Number; unit: participants
Arm/Group | Stratum 2
Number analyzed (Participants) | 12
participants | 12

3. Primary Outcome: Toxicity
Description: Number of participants experiencing adverse events
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Population: All evaluable participants for Stratum 1 and 2 combined.
Measure: Number; unit: Participants
Groups:
- Stratum 1: Patients ≥ 3 years old with progressive plexiform neurofibroma(s) with the potential to cause significant morbidity.
- Stratum 2: Patients ≥ 3 years old and plexiform neurofibroma(s) without documented radiographic progression at trial entry. The endpoint will be radiographic response.
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 49 | 13
Participants | 49 | 13

4. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus Administered to This Patient Population (Clearance Liters/Hour (L/h))
Description: An iterative 2-stage Bayesian method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Pediatric Patients (3 through 18) with Neurofibromatosis Type 1 - Clearance liters/hour (L/h). Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: Clearance liters/hour (L/h)
Groups:
- Stratum 1: Design
  • Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing.
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
Clearance liters/hour (L/h) | 11.8 (4.6)

5. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus When Administered to This Patient Population Using Liters/Hour Per Population Median Weight of 70kg (L/h70kg)
Description: An iterative 2-stage Bayesian method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Stratum 1 used allometrically scaled clearance (clearance scaled to a 70kg individual). Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: L/h/70kg
Groups:
- Stratum 1: Design
  • Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing. Sirolimus, Rapamycin: This phase II study will evaluate children and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with sirolimus. It is divided in two strata. The first stratum will evaluate time to progression (TTP) in children and adults with NF1 and progressive plexiform neurofibromas with the potential to cause sign
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
L/h/70kg | 23.7 (6.7)

6. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus When Administered to This Patient Population - (Clearance (L/h Per 1.85 m^2)
Description: An iterative 2-stage Bayesian Method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Stratum 1, Neurofibromatosis Type 1 Patients Clearance (L/h per 1.85 m^2). Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: L/h per 1.85 m^2
Groups:
- Stratum 1: Design
  • Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing.
  Sirolimus, Rapamycin: This phase II study will evaluate children and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with sirolimus. It is divided in two strata. The first stratum will evaluate time to progression (TTP) in children and adults with NF1 and progressive plexiform neurofibromas with the potential to cause significant morbidity treated with sirolimus. The second stratum will evaluate objective radiographic response to sirolimus in children and adults with NF1 and inoperable plexiform neurofibromas with the potential to cause significant morbidity that do not have documented progression of the PN at time of trial entry.
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
L/h per 1.85 m^2 | 6.4 (2.5)

7. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus When Administered to This Patient Population- Therapeutic Dose (mg/m^2 Per Dose)
Description: An iterative 2-stage Bayesian Method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Stratum 1, Neurofibromatosis Type 1 patients - Therapeutic Dose (mg/m^2 per dose). Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: Therapeutic Dose mg/m^2 per dose
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
Therapeutic Dose mg/m^2 per dose | 2.0 (0.7)

8. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus in When Administered to This Patient Population - Therapeutic Dose (mg/kg Per Dose)
Description: An iterative 2-stage Bayesian Method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Stratum 1, Neurofibromatosis Type 1 patients (Ages 3 to 18) Therapeutic Dose (mg/kg per dose). Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: Therapeutic Dose (mg/kg per dose)
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
Therapeutic Dose (mg/kg per dose) | 0.08 (0.04)

9. Primary Outcome: To Characterize the Pharmacokinetic Profile of Sirolimus When Administered to This Patient Population - Therapeutic Dose (mg/kg)^0.75
Description: An iterative 2-stage Bayesian method was used for the PK parameter analyses
Time Frame: Pre-dose; Day 1 at 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 10.0 to 12.0 hours
Population: Stratum 1, Neurofibromatosis Type 1 patients (ages 3 to 18) - Therapeutic Dose (mg/kg)^0.75. Stratum 2 did not meet the 6 month response criteria; therefore, was not analyzed for pharmacokinetic profiles.
Measure: Mean (Standard Deviation); unit: Therapeutic Dose (mg/kg)^0.75
Arm/Group | Stratum 1
Number analyzed (Participants) | 44
Therapeutic Dose (mg/kg)^0.75 | 0.14 (0.05)

10. Secondary Outcome: To Evaluate the Quality of Life During Treatment With Sirolimus by Assessing Preliminary Correlations of Response With Quality-of-life Outcomes
Description: Self-reported, age-appropriate PedsQL Scale. Assessments included: Inventory for physical function, emotional function, social function and school function - number system 0-4 was used with 4 being the worse maximum threshold); inventory for chronic illness used a 5-point likert scale - 5 being the worst maximum threshold; Skindex-Teen used a scale of 0 to 100 - the higher the number the more frequent the experience; Pain intensity was measured using a line with a happy and sad face - marks toward the sad face indicated more intense pain; and, the McGill Pain Questionnaire - higher values indicating worse pain of a scale from 0-3. All assessments were combined for an overall PedsQL score by rating each item 0-4, then reverse transforming each to a 0 - 100 scale. The total scores were calculated by averaging the item scores, with higher scores being better.
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Population: Stratum 1 patients with Neurofibromatosis Type 1; all ages - Change from Baseline to Course 3. Stratum 2 did not meet the requirements for response at the 6 month time point. Therefore, Stratum 2 was not analyzed for this aim.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stratum 1
Number analyzed (Participants) | 23
Units on a scale | 2.8 (9.59)

11. Secondary Outcome: To Assess the Value of Three-dimensional MRI (3-D MRI) in the Evaluation of Plexiform Neurofibromas and Paraspinal Neurofibromas, and to Compare 3-D MRI to Conventional Two-dimensional MRI (2-D MRI) and One Dimensional MRI (1-D MRI) Data Analysis
Description: The study provided central review of all MRIs using a three-dimensional volumetric protocol. As the STOPN protocol began, research had already demonstrated the superiority of this approach to 1-D or 2-D analyses, so these were not used in the STOPN study.
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Population: The data for this outcome wasn't collected because prior to the study, it was determined that MRI (3-D MRI) was already superior, so the MRI was not performed on any of the participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: To Asses Preliminary Correlations of Radiographic Response With Changes in Pharmacodynamics Parameters Including p70s6 Kinase Activity in Peripheral Blood Mononuclear Cells.
Description: Response by Volumetric MRI.
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Population: Samples were inadequate in quantity to allow for this analysis.
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: To Evaluate the Effect of Sirolimus on Clinical Response by Reduction in Pain, or Improvement in Function or Performance Scale.
Description: There were no data collected for this outcome measure.
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: To Evaluate Pharmacogenetic Polymorphisms of Cytochrome P450 3A4 & 3A5 Alleles and P-glycoprotein/MDR for Their Influence on the Metabolism of Sirolimus in This Patient Population.
Description: Trough concentration of sirolimus is reported in nanograms per mL.
Time Frame: 24 weeks Stratum 1 Only
Population: Subjects in Stratum 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 37 | 0
ng/mL | 9.37 (2.48) |

15. Secondary Outcome: To Evaluate the Role of Apolipoprotein E Genotypes as Predictors for Development of Hyperlipidemia During Therapy With Sirolimus.
Description: Number of patients who experienced hyperlipidemia is being reported.
Time Frame: 24 weeks Stratum 1 / 48 weeks Stratum 2
Measure: Number; unit: participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 46 | 12
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Description: Stratum 1
Groups:
- Stratum 1: Non-randomized, single arm interventional strata for inoperable Plexiform Neurofibromas with potential to cause significant morbidity with evidence of progression.
  Sirolimus oral solution will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment course) with pharmacokinetically-guided dosing. Disease status will be evaluated using volumetric MRI analysis at regular intervals.
Arm/Group | Stratum 1 | Stratum 2
Serious Adverse Events (participants affected / at risk) | 20/46 | 4/12
Other Adverse Events (participants affected / at risk) | 8/46 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=46) | Stratum 2 (N=12)
Vomiting/Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Infection - Viral (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
ALT, AST & GGP (Investigations) | 1 (1) | 0 (0) — Grade 3
Fever due to infection - Viral (Infections and infestations) | 1 (1) | 0 (0) — Grade 3
Local Complication - Device/Prosthesis (Eye) (Surgical and medical procedures) | 1 (1) | 0 (0) — Grade 3
Infection with Normal ANC (Pneumonia) (Infections and infestations) | 1 (1) | 0 (0) — Grade 3
Left Ventricular Systolic Dysfuntion (Grade1) with Admission (Grade 2) (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2
Pain (General disorders) | 1 (1) | 0 (0) — Grade 3
Motor Neuropathy - Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) — Grade 4
Infection - UTI (Normal ANC) (Infections and infestations) | 1 (1) | 0 (0) — Grade 3
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 4
NF1 Related Planned Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Left Distal Femur and Left Proximal Tibid Epiphysiodesis (Unrelated to drug) Grade 3
Surgery - Injury to the Musculoskeletal (Lower Extremity) (Surgical and medical procedures) | 1 (1) | 0 (0) — Grade 3
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
Altered Mental State (Nervous system disorders) | 1 (1) | 0 (0) — Grade 2
Strep Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 3
Influenza Virus Type B (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
Pain - ABD and Leg (General disorders) | 1 (1) | 0 (0) — Grade 2
AST (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3
ALT (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3
Hydroureteronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) — Resulting in Increased Creatinine - Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=46) | Stratum 2 (N=12)
Headache (Nervous system disorders) | 2 (2) | 1 (1) — Grade 2
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) — Grade 2
Low ANC (Investigations) | 1 (1) | 0 (0) — Grade 2
Low WBC (Investigations) | 1 (1) | 0 (0) — Grade 2
Pain - Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Low Leukocytes (Investigations) | 1 (1) | 0 (0) — Grade 2
Stomatitis/Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1
Neutropenia (Investigations) | 1 (1) | 0 (0) — Grade 2
Neutropoenia (Investigations) | 4 (4) | 0 (0) — Grade 2
Mucositis (Gastrointestinal disorders) | 8 (8) | 2 (2) — Grade 2
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0) — Grade 3
Lymphopenia (Investigations) | 4 (4) | 0 (0) — Grade 2
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Grade 2
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Mouth Sores (Gastrointestinal disorders) | 4 (4) | 2 (2) — Grade 2
Weight Loss (Investigations) | 1 (1) | 0 (0) — Grade 2
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2
Pain -- Adominal (Gastrointestinal disorders) | 3 (3) | 3 (3) — Grade 2
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Grade 2
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) — Grade 2
Hypercholesteremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2
Fatigue (General disorders) | 3 (3) | 0 (0) — Grade 2
Fever (General disorders) | 4 (4) | 1 (1) — Grade 2
Mood Alteration (Psychiatric disorders) | 2 (2) | 0 (0) — Grade 2
ALT (Investigations) | 1 (1) | 1 (1) — Grade 3
AST (Investigations) | 1 (1) | 0 (0) — Grade 3
GGT (Investigations) | 1 (1) | 0 (0) — Grade 3
WBC (Investigations) | 1 (1) | 0 (0) — Grade 2
Lukopenia (Investigations) | 1 (1) | 1 (1) — Grade 2
Neutropenia (Investigations) | 2 (2) | 0 (0) — Grade 3
Allergic Reaction - Bactrim (Immune system disorders) | 1 (1) | 0 (0) — Grade 2
Hirsutism several locations (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Legs, Trunk, Back and Face Grade 2
New Neurofibroma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — NF on Back - Grade 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) — Grade 2
Infection with Normal ANC - Lung (Infections and infestations) | 1 (1) | 0 (0) — Pneumo Grade 3
Mood Alteration - Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 3
Infection -Derm/Skin (Infections and infestations) | 1 (1) | 0 (0) — Cellulitis Grade 2
Infection w/ Normal ANC (Infections and infestations) | 2 (2) | 0 (0) — Grade 2
Infection w/ Normal ANC: Otitis Media (Infections and infestations) | 1 (1) | 0 (0) — Grade 3
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 2
Leukocytes (Investigations) | 1 (1) | 0 (0) — Grade 2
Neutrophils (Investigations) | 5 (5) | 1 (1) — Grade 2
Pain - Throat (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Neutrophils (Investigations) | 2 (2) | 0 (0) — Grade 3
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
ARDS (Secondary to RSV) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 4
Triglycerides - Serum High (Metabolism and nutrition disorders) | 2 (2) | 0 — Grade 2
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Grade 2
LDL Cholesterol 235MG/DL (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3
Total Cholesterol (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 2
Neutrophils/Granulocytes (ANC/AGC) (Investigations) | 4 (4) | 0 (0) — Grade 2
Infection - Upper Airway NOS (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
Neutrophils/Granulocytes Low (Investigations) | 1 (1) | 0 (0) — Grade 3
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
Otitis - Middle Ear (Infections and infestations) | 2 (2) | 0 (0) — Grade 2
Pain - Leg (General disorders) | 1 (1) | 0 (0) — Grade 2
Febrile Neutropenia (Investigations) | 1 (1) | 0 (0) — Grade 3
Infection - Ear (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
Face Tenderness/Swollen/Headaches/Aches (Nervous system disorders) | 0 (0) | 1 (1) — Grade 2
AST (Investigations) | 0 (0) | 1 (1) — Grade 2
Infection - fever of unknown temperature / Cold (Infections and infestations) | 0 (0) | 1 (1) — Grade 2
High Blood Pressure (Vascular disorders) | 0 (0) | 1 (1) — Grade 2
Mouth Sore - Upper Inner Left Corner (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2
Edema - Knee Swelling (General disorders) | 0 (0) | 1 (1) — Grade 2
Pain - Knee (General disorders) | 0 (0) | 1 (1) — Grade 2
Low Hemoglobin Delaying Start of Cycle (Investigations) | 0 (0) | 1 (1) — Grade 2
Infection - Thrush w/OK ANC (Infections and infestations) | 0 (0) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No